Official Title of the Study:

A Randomized Controlled Study Investigating the Effectiveness of Intravenous Dexamethasone Prophylaxis in Preventing Post-operative Urinary Retention in Spinal Anesthesia at Al-Makassed Hospital

**NCT Number: NCT07077850** 

Date of Document: 01/07/2025

| REC OFFICE USE | |
|---------------------------------------|-----------------------|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
| Date Received | |
| Institute/Centre/Faculty | titute/Centre/Faculty |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |



Ethics Research Committee, Al-Quds University

### 1. Project Title (in full)

Effectiveness of Intravenous Dexamethasone Prophylaxis in Preventing Post-operative Urinary Retention in Spinal Anaesthesia at Al-Makassed Hospital

### **RESEARCH PERSONNEL**

#### **General Supervisor**

| Name | Dr. Mohammed Maree |
|---|---|
| Title | General surgeon |
| Qualifications | MD |
| University Position Held: employee, affiliate (indicate type; eg. honorary associate, clinical academic), visiting Full mailing address | clinical academic Faculty of Medicine Al-Quds University Ramallah, Palestine |
| Telephone | 00972592309896 |
| Fax | - |
| E-mail | mohammedmaree1983@gmail.com |

#### **Principal Investigator**

| Name | Dr. Abeer Dar Hasan |
|----------------|---------------------------|
| Title | Resident doctor – surgery |
| Qualifications | MD |

| REC OFFICE USE | |
|---------------------------------------|------------------------|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
| Date Received | |
| Institute/Centre/Faculty | stitute/Centre/Faculty |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |



## Research Ethics committee (REC)

### Application Form

Ethics Research Committee, Al-Quds University

| University Position Held:<br>employee, affiliate (indicate<br>type; eg. honorary associate,<br>clinical academic), visiting | - |
|---|---|
| Full mailing address | Jerusalem, Palestine |
| Telephone | 00972534541877 |
| Fax | - |
| E-mail | abee.9.1994@gmail.com |

### Associate Investigator(s)

| Associate Investigator 1 | |
|---|---|
| Name | Dr. Ahlam Hammoudeh |
| Title | Resident doctor – anesthesia |
| Qualifications | MD |
| University Position Held:<br>employee, affiliate (indicate<br>type eg honorary associate,<br>clinical academic), visiting | - |
| Full mailing address | Jerusalem , Palestine |
| Telephone | 00972595744577 |
| Fax | - |
| E-mail | ahlamhammoudeh123@yahoo.com |

| Associate Investigator 2 | |
|--------------------------|------------------------------|
| Name | Dr. Islam Khairaldin |
| Title | Resident doctor – anesthesia |
| Qualifications | MD |

| REC OFFICE USE | |
|---------------------------------------|----------------------|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
| Date Received | |
| Institute/Centre/Faculty | |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |



## Research Ethics committee (REC)

### Application Form

| University Position Held:<br>employee, affiliate (indicate<br>type eg honorary associate,<br>clinical academic), visiting | - |
|---|---|
| Full mailing address | Jerusalem , Palestine |
| Telephone | 00972533491136 |
| Fax | - |
| E-mail | islamkhairaldeen@gmail.com |

| Associate Investigator 3 | |
|---|---|
| Name | Dr. Majdi Abu Daoud |
| Title | Resident doctor – surgery |
| Qualifications | MD |
| University Position Held:<br>employee, affiliate (indicate<br>type eg honorary associate,<br>clinical academic), visiting | - |
| Full mailing address | Bethlehem, Palestine |
| Telephone | 00972595414606 |
| Fax | - |
| E-mail | majdi.aziz1998@gmail.com |

| Associate Investigator 4 | |
|---|---|
| Name | Dr. Mohammad Qino |
| Title | Resident doctor – surgery |
| Qualifications | MD |
| University Position Held:<br>employee, affiliate (indicate<br>type eg honorary associate,<br>clinical academic), visiting | - |
| Full mailing address | Jerusalem, Palestine |

| REC OFFICE USE | |
|---------------------------------------|-----------------------|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
| Date Received | |
| Institute/Centre/Faculty | titute/Centre/Faculty |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |



## Research Ethics committee (REC)

### Application Form

| Telephone | 00972597484208 |
|-----------|-------------------|
| Fax | - |
| E-mail | M.qinoo@gmail.com |

| Associate Investigator 5 | |
|---|---|
| Name | Anas Barabrah |
| Title | Medical Student |
| Qualifications | undergraduate |
| University Position Held:<br>employee, affiliate (indicate<br>type eg honorary associate,<br>clinical academic), visiting | Medical Student Faculty of Medicine Al-Quds University |
| Full mailing address | Ramallah, Palestine |
| Telephone | 0597159258 |
| Fax | - |
| E-mail | anasmufeed3@gmail.com |

| Associate Investigator 6 | |
|---|---|
| Name | Tareq Jarrar |
| Title | Medical Student |
| Qualifications | undergraduate |
| University Position Held:<br>employee, affiliate (indicate<br>type eg honorary associate,<br>clinical academic), visiting | Medical Student Faculty of Medicine Al-Quds University |
| Full mailing address | Ramallah, Palestine |
| Telephone | 00972595076137 |
| Fax | - |
| E-mail | tareq.jarrar2@students.alquds.edu |

| REC OFFICE USE | |
|---------------------------------------|----------------------|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
| Date Received | |
| Institute/Centre/Faculty | |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |



| Associate Investigator 7 | |
|---|---|
| Name | Amani Ahmed |
| Title | Resident doctor-Surgery |
| Qualifications | MD |
| University Position Held:<br>employee, affiliate (indicate<br>type eg honorary associate,<br>clinical academic), visiting | - |
| Full mailing address | Jerico, Palestine |
| Telephone | 00972569045086 |
| Fax | - |
| E-mail | amanibashar243@gmail.com |

| Associate Investigator 8 | |
|---|---|
| Name | Osama Mohammed Sawalha |
| Title | MD |
| Qualifications | Anaesthesiologist |
| University Position Held:<br>employee, affiliate (indicate<br>type eg honorary associate,<br>clinical academic), visiting | - |
| Full mailing address | Tulkarem , Palestine |
| Telephone | 00972598603554 |
| Fax | • |
| E-mail | modosawalhair@gmail.com |

| Associate Investigator 9 | |
|--------------------------|-----------------------|
| Name | Khaled Nassed Alshawa |
| Title | MD ,MRCS |

| REC OFFICE USE | |
|---------------------------------------|----------------------|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
| Date Received | |
| Institute/Centre/Faculty | |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |



#### Research Ethics committee (REC)

#### **Application Form**

Ethics Research Committee, Al-Quds University

| Qualifications | General Surgeon |
|---|---|
| University Position Held:<br>employee, affiliate (indicate<br>type eg honorary associate,<br>clinical academic), visiting | Clinical Lecturer Faculty of medicine Azhar University |
| Full mailing address | Gaza, Palestine |
| Telephone | 00972599335031 |
| Fax | - |
| E-mail | khaledshawa@gmail.com |

#### **PROJECT AND SITE DETAILS**

2. Please provide details of the research setting (Research laboratory, Hospital, etc)

This research project will be done at Al-Makassed Hospital by surgery, anaesthesia doctors, and undergraduate medical students. Data will be collected verbally in the surgery department by resident doctors.

3. Provide information to demonstrate that the researchers involved in the project have the necessary training, expertise and experience to carry out their role in the research.

This research will be supervised by Dr. Mohammad Maree and sponsored by AMRA. All authors had enrolled in previous similar research projects. Most of the research team completed the following modules from TRREE:

Module 1: Introduction to Research Ethics

Module 3: Informed Consent Module 3.2: Good Clinical Practice

4. Please outline (or attach) the proposed procedure for dealing with any health emergencies that may arise during the conduct of the research. If the Principal Investigator at the proposed University site is

| REC OFFICE USE | |
|---------------------------------------|----------------------|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
| Date Received | |
| Institute/Centre/Faculty | |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |



## Research Ethics committee (REC)

#### Application Form

Ethics Research Committee, Al-Quds University

not a health practitioner, please provide details of the medical practitioner who will be responsible for

| | dealing with medical emergencies. | | |
|---|---|---|---|
| | | | of general surgery specialists and well-trained doctors. Therefore, if any emergency research process, they will deal with it. |
| 5. | Risk as | ssessme | ent (please indicate that the following are accurate): |
| | The site has adequate data protection and security systems to ensure protection of participan privacy | | |
| | <b>√</b> | ☑ The site has adequate, secure systems for storage of investigational products | |
| | V | Partici | pants are able to report adverse events and study outcomes reliably |
| 6. | 6. Is this research at the University site commercially sponsored? | | |
| | | <b>√</b> | NO |
| | | | YES – please provide a copy of the certificates |

| REC OFFICE USE | |
|---------------------------------------|----------------------|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
| Date Received | |
| Institute/Centre/Faculty | |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |



Research Ethics committee (REC)

Application Form

Ethics Research Committee, Al-Quds University

**DECLARATION BY INVESTIGATORS** 

I confirm that I have read and understand the attached Code of Good Practise and Helsinki declaration in Research Conduct in Human Research.

I confirm that I have read and understand the Code of Good Practise and Helsinki declaration in Research Conduct in Human (Provided and declared by the Ethics Research Committee, Al-Quds University)

I confirm that the above information is accurate, and that the project will continue in accordance with the Human Research Ethics Committee approved protocol.

| General Supervisor | Dr.Mohammed Maree<br>General &laparoscopic Surgeon | |
|---|---|---|
| Dr. Mohammed Maree | | 10/02/202 |
| Name | Signature | Date |
| Principal Investigator | 24 | |
| Dr. Abeer Dar Hasan | | 10/02/202 |
| Name | Signature | Date |
| Associate Investigator(s) | -092 (NO) | |
| Dr. Ahlam Hammoudeh | Control of the second of the s | _10/02/202 |
| Name | Signature | Date |
| Dr. Islam Khairaldin | | 10/02/202 |
| Name | Signature | Date |
| Dr. Majdi Abu Daoud | OR MASOE A | 10/02/202 |
| Name | Signature | Date |
| | Up | 10/02/202 |

| REC OFFICE USE | |
|---------------------------------------|----------------------|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
| Date Received | |
| Institute/Centre/Faculty | |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |



## Research Ethics committee (REC)

### Application Form

| Dr. Mohammad Qino | • | |
|---------------------|-----------|------------|
| Name | Signature | Date |
| Anas Barabrah | | _10/02/202 |
| Name | Signature | Date |
| Tareq Jarrar | | 10/02/202 |
| Name | Signature | Date |
| A : Al I | S. Lua | 10/06/202 |
| Amani Ahmed<br>Name | Signature | Date |
| Osama Sawalha | Laur | 10/02/202 |
| Name | Signature | Date |
| | | 10/02/202 |
| Khaled Alshawa Name | Signature | Date |
| IVAIIIO | Signature | Daio |

| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
|---|---|
| Date Received | |
| Institute/Centre/Faculty | |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |
| TO THE PARTY OF TH | |
| Al-Quds University | |
| Al-Quds University Research Ethics com | mittee (REC) |
| Al-Quds University Research Ethics com Application Form | mittee (REC) |
| Research Ethics com<br>Application Form | |
| Research Ethics com | |

| The e | thics | committee of Al-Makassed Hospital |
|---|---|---|
| 1.3 | (a) | Indicate the proposed date of commencement of the project. Projects should not commence without the prior written approval of the REC. |
| Date | July | 2025 |
| | | (b) Indicate the proposed completion date of the project. |
| Date | Jan 2 | 2026 |

1.4 (a) Has this protocol received research funding/contracting or is this submission being made as part of an application for research funding/contracting?

N
Y

If you answered YES, list the funding/contracting bodies to which you have submitted, or intend to submit, this project. Attach a copy of the grant application(s), contract(s) or similar agreement(s).

| REC OFFICE USE | |
|---------------------------------------|----------------------|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
| Date Received | |
| Institute/Centre/Faculty | |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |



## Research Ethics committee (REC)

Application Form

| , pp. oad on to the |
|-----------------------------------------------|
| Ethics Research Committee, Al-Quds University |
| Funding/Contracting body 1: |
| Funding/Contracting body 2: |
| Funding/Contracting body 3: |

## SECTION 2: NATURE OF RESEARCH

| 2.1 | The nature of this project is most appropriately described as research involving: (more than one may apply): | |
|---|---|---|
| _ | behavioural observation | |
| _ | self-report questionnaire(s) | Y 🔽 |
| _ | interview(s) | Υ |
| _ | qualitative methodologies (e.g. focus groups) | Y 🔽 |
| _ | psychological experiments | Y |
| _ | epidemiological studies | Y |
| _ | data linkage studies | Υ |
| _ | psychiatric or clinical psychology studies | Υ |
| _ | human physiological investigation(s) | Υ |

| REC OFFICE USE | |
|---------------------------------------|----------------------|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
| Date Received | |
| Institute/Centre/Faculty | |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |



Ethics Research Committee, Al-Quds University

- biomechanical device(s)
- human tissue
- human genetic analysis
- a clinical trial of drug(s) or device(s)
- Other (please specify in the box below)

Proceed to Section 3.

| REC OFFICE USE | |
|---------------------------------------|----------------------|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
| Date Received | |
| Institute/Centre/Faculty | |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |



Ethics Research Committee, Al-Quds University

**SECTION 3: PARTICIPANTS AND RECRUITMENT** 

| 3.1 | (a) | What is the age range of all participants involved in this study? |
|---|---|---|
| | () | , |

| ≥ 18 (Adult | s) | | |
|---|---|---|---|
| (b) | Are the participants include children (defined by statute for this purpose as anyone under 18) | Y | V<br>N |

If you answered NO, give reasons why not.

Post-operative urinary retention might be a relatively rare occurrence in children compared to adults. Also, agerelated differences in etiology, risk factors, and management of postoperative urinary retention might differ between adults and children due to anatomical, physiological, and developmental variations.

#### 3.2 Are the participants:- (more than one may apply)

| - | in a teacher-student relationship with the researchers or their associates? | |
|---|---|---|
| - | in an employer-employee relationship with the researchers or their associates? | |
| - | in any other dependent relationship with the researchers or their associates? | I V |
| _ | prisoners? | Y V |
| _ | refugees? | Ĭ |
| _ | members of the security services? | Ť |

| REC OFFICE USE | | | | |
|---|---|---|---|---|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | | | | |
| Date Received | | | | |
| Institute/Centre/Faculty | | | | |
| Campus | | | | |
| | Master's project | | | |
| | Grants Awarded | | | |
| | Small Grants Awarded General | | | |
| | Clinical Trials | | | |
| <ul><li>in a doctor-<br/>with the res</li></ul> | tee, Al-Quds University | | Y<br>Y<br>Y<br>Y<br>V | ] |
| , | | | | |
| | sample size for the study? Co to be achieved. | omment on how this sample size w | ill allow the aims | S |
| | significance level. This allows fo | le size was calculated by a power an | | |
| 3.4 Will participants re | eceive any reimbursement | | | |
| | socied any reminaraement | | N Y | Y |
| | | | 19 1 | • |
| If you answered YE | S, what is the amount or nature | e of the reward and the justification fo | or this? | |

| DEC | OFFICE USE | | | 1 |
|---|---|---|---|---|
| HUM | AN RESEARCH<br>CS COMMITTEE No | | | |
| | Received | | | |
| | | _ | | |
| | tute/Centre/Faculty | | | |
| Cam | pus | M4 | 1 | |
| | | Master's project Grants Awarded | | |
| | | Small Grants Awarded | | |
| | | General | | |
| | | Clinical Trials | | |
| Res<br>App<br>Ethic | Quds University earch Ethics com lication Form es Research Commit eeed to section 4 | <b>mittee (REC)</b><br>tee, Al-Quds University | | |
| SEC | SECTION 4: PRIVACY | | | |
| 4.1 | personal nature (consent? | either identifiable or po | otentia | dentify, collect, use, or disclose information of a ally identifiable) about individuals without their V N Y De sought and how many records will be accessed. |
| IF YO | U ANSWERED NO,<br>5 | YOU DO NOT NEED TO | о сом | PLETE ANY MORE OF SECTION 4. GO TO SECTION |
| Plea | se provide details | | | |

Proceed to Section 5.

SECTION 5: COLLECTION OF DATA

| REC OFFICE U | JSE | |
|---|---|---|
| HUMAN RESE | | |
| Date Received | | |
| Institute/Centr | e/Faculty | |
| Campus | | |
| - | | Master's project |
| | | Grants Awarded |
| | | Small Grants Awarded |
| | | General |
| | | Clinical Trials |
| Al-Quds University Research Ethics committee (REC) Application Form | | |
| Etnics Reseal | cn Committ | ee, Al-Quds University |
| or othe | 5.1 Will any part of the study involve recordings using audio tape, film/video, or other electronic medium? If you answered YES, what is the medium and how it will be used? | |
| 5.2 Does your research involve the <u>secretive</u> use of photographs, tape-recordings, or any other form of record-taking? N Y | | |
| If you answered YES, provide details and a justification for the secrecy. | | |

5.3 (a) How will the results of the study be disseminated (e.g. via publication in journals and presentations in scientific meetings)?

The results will be published in a journal, and shared in conferences.

5.4 How will the confidentiality of the data, including the identity of participants, be ensured during collection and dissemination?

| REC OFFICE USE | |
|---------------------------------------|----------------------|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
| Date Received | |
| Institute/Centre/Faculty | |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |



Ethics Research Committee, Al-Quds University

| 5.5 | (a) | (a) What is the proposed storage location of, and access to, materials collected during the study (including files, audiotapes, questionnaires, videotapes, photographs)? | | |
|---|---|---|---|---|
| | | Please cross (X) the appropriate box: Principal investigator's Office Faculty / Departmental Office Other (Please provide details below) | Room No.<br>Room No. | Building Building |
| A shared Google drive by authors | | | | |
| | (b) | On completion of the study, where will the (including files, audiotapes, questionnaires, Please cross (X) the appropriate box: | | |
| | | Principal Investigator's Office Faculty / Departmental Office Other (Please provide details below) | Room No.<br>Room No. | Building Building |
| | | A shared Google drive by authors | | |

Participants will be asked some questions after the surgery, no collection of their name or address will be done.
Participants' file number will not be shared with the data or the research results.

| REC OFFICE USE | |
|---------------------------------------|----------------------|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
| Date Received | |
| Institute/Centre/Faculty | |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |



| Passayah Ethias sammittas (BEC) | |
|---|---|
| Research Ethics committee (REC) Application Form | |
| Ethics Research Committee, Al-Quds University | |
| SECTION 6: ASSESSMENT OF RISKS | |
| 6.1 Indicate if the participants might experience any of the following: | |
| Risk of physical harm (e.g., falling, muscle pain) | |
| Y Physical discomfort (e.g., tiredness, weakness, nausea) Y | <u> </u> |
| Risk of psychological or emotional harm (e.g., trauma) Y | |
| Psychological or emotional discomfort (e.g., anxiety, stress, loss of confidence, regret for disclosing information) | personal |
| Υ | |
| Legal repercussions for participating in the study (e.g., possibility of being sued, charged with crimin Y | al activity) |
| 6.2 POTENTIAL RISK TO PARTICIPANTS AND RISK MANAGEMENT PROCEDURES Identify, as far as possible, all potential risks to participants (e.g. physical, psychological, se economic), associated with the proposed research. Please explain what risk management probe put in place. | |
| <ul> <li>No potential risks.</li> <li>Any patient who is expected to develop drug-related complications will be excluded from t study.</li> </ul> | the |

6.3 ARE THERE ANY SPECIFIC RISKS TO RESEARCHERS THAT ARE GREATER THAN THOSE ENCOUNTERED IN NORMAL DAY TO DAY LIFE?

| REC OFFICE USE | |
|---------------------------------------|----------------------|
| HUMAN RESEARCH<br>ETHICS COMMITTEE No | |
| Date Received | |
| Institute/Centre/Faculty | |
| Campus | |
| | Master's project |
| | Grants Awarded |
| | Small Grants Awarded |
| | General |
| | Clinical Trials |



Ethics Research Committee, Al-Quds University

| YES | V | NO | (If YES, please describe.) |
|-----|---|----|----------------------------|

End of the application